CLINICAL TRIAL: NCT04937517
Title: The Role of the Apex of the Deep Cartilage in Assessing Femoral Tunnel Position for Anterior Cruciate Ligament Reconstruction
Brief Title: ADC in Assessing Femoral Tunnel Position
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ADC
Record Dates: First submitted 2021-06-16; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: ACL Injury
Keywords: femoral tunnel; apex of the deep cartilage（ADC）
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To examine the consistency between postoperative CT scan and intraoperative arthroscopic measurement in evaluating femoral tunnel position for anterior cruciate ligament （ACL）reconstruction，both using the apex of the deep cartilage（ADC）as the marker.

DETAILED DESCRIPTION:
The position of the center of femoral tunnel was decided in the complete femoral stub. Then the length from the ADC to the anterior cartilage margin（L1）and to the center of femoral tunnel（l1），as well as the center to the distal cartilage margin（D1）were measured under arthroscopy and on post-operative CT scan（L2，l2 and D2）. Moreover，P1 and P2 were calculated through l1/L1 and l2/L2.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-55 who need anterior cruciate ligament reconstruction

Exclusion Criteria:

* Volunteers unsuitable for anterior cruciate ligament reconstruction

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults aged 18-55 who need and suitable anterior cruciate ligament reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
length from ADC to anterior cartilage margin (L1) under arthroscopy | during operation
  length from ADC to anterior cartilage margin (L1) under arthroscopy
length from ADC to the center of femoral tunnel (l1) under arthroscopy | during operation
  length from ADC to the center of femoral tunnel (l1) under arthroscopy
length from the center of femoral tunnel to the distal cartilage margin(D1) under arthroscopy | during operation
  length from the center of femoral tunnel to the distal cartilage margin(D1) under arthroscopy
length from ADC to anterior cartilage margin (L2) on CT | 1 day after operation
  length from ADC to anterior cartilage margin (L2) on CT
length from ADC to the center of femoral tunnel (l1) on CT | 1 day after operation
  length from ADC to the center of femoral tunnel (l1) on CT
length from the center of femoral tunnel to the distal cartilage margin(D1) on CT | 1 day after operation
  length from the center of femoral tunnel to the distal cartilage margin(D1) on CT

CONTACTS AND LOCATIONS:
Locations (1):
- Ma Yong, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Publication of academic papers

REFERENCES:
- [Background] Hofbauer M, Muller B, Murawski CD, van Eck CF, Fu FH. The concept of individualized anatomic anterior cruciate ligament (ACL) reconstruction. Knee Surg Sports Traumatol Arthrosc. 2014 May;22(5):979-86. doi: 10.1007/s00167-013-2562-4. Epub 2013 Jun 6. PMID 23740328
- [Background] Inderhaug E, Larsen A, Strand T, Waaler PA, Solheim E. The effect of feedback from post-operative 3D CT on placement of femoral tunnels in single-bundle anatomic ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2016 Jan;24(1):154-60. doi: 10.1007/s00167-014-3355-0. Epub 2014 Oct 2. PMID 25274095
- [Background] Hart A, Han Y, Martineau PA. The Apex of the Deep Cartilage: A Landmark and New Technique to Help Identify Femoral Tunnel Placement in Anterior Cruciate Ligament Reconstruction. Arthroscopy. 2015 Sep;31(9):1777-83. doi: 10.1016/j.arthro.2015.03.026. Epub 2015 May 15. PMID 25980920
- [Derived] Shi W, Zhang J, Meng Q, Chen N, Shen Q, Li S, Cao Z, Ao Y, Ma Y. The apex of the deep cartilage is a stable landmark to evaluate the femoral tunnel position in ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2023 Jan;31(1):256-263. doi: 10.1007/s00167-022-07090-4. Epub 2022 Aug 13. PMID 35962841